CLINICAL TRIAL: NCT06604403
Title: Effect of Massage Applied to Hemodialysis Patients on Comfort Level and Fatigue
Brief Title: Effectiveness of Massage Applied to Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Yildirim (Other)
Responsible Party: Sponsor-Investigator, Zeynep Yildirim, Research Assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Massage
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nurse's Role
Keywords: Massage; Hemodialysis Patients; Nursing; Comfort; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Massage Group (Experimental): Patients in the intervention group will receive post-hemodialysis massage twice a week for four weeks.
  Interventions: Other: Massage
- Control Group (No Intervention): Routine nursing care was given to the patients in this group without any message.

INTERVENTIONS:
Other: Massage — After the hemodialysis, the patients will receive a 15-20 minute hand and foot massage. This application will be applied to the patients in two weekly dialysis sessions for a total of 8 sessions for four weeks. Before starting the massage applications, the patient's hands and feet will be washed and dried thoroughly. The patients will be given a semi-sitting or lying position that they can feel comfortable in. Before starting the hand and foot massage, the researcher will gently rub and warm their hands and wrists. The massages will start with a hand massage. A foot massage will be performed after the hand massage. 3-5 drops of baby oil applied at room temperature will be used to reduce friction during the massage. Effleurage, petrissage and friction styles of the massage will be applied.
  Arms: Massage Group

SUMMARY:
This study was conducted to determine the effect of massage on comfort and fatigue levels of hemodialysis patients.

DETAILED DESCRIPTION:
Chronic renal failure (CRF) is a health problem that causes significant mortality and morbidity worldwide. The prevalence of the disease is increasing worldwide, especially in developing countries. Hemodialysis (HD) is the most common treatment method for CRF in the world. Approximately 90% of patients with CRF receive HD treatment. Despite advances in technology and medical care due to HD treatment, patients experience many physical and psychosocial symptoms. It is emphasized that comfort is significantly negatively affected in HD patients due to reasons such as the direct impact of HD treatment on the daily and social lives of patients. Increasing the comfort level is important for the patient to continue their daily life activities. In addition, comfort is accepted as the basis of quality nursing care. Increasing the comfort levels of HD patients provides lower comorbidity and mortality rates and improvement in institutional patient outcomes. Fatigue, one of the physical symptoms seen in HD patients, affects 60-95% of patients. Fatigue increases the patients' dependency levels, reduces their physical capabilities, negatively affects the patient and their family economically and reduces their quality of life. Therefore, effective management of fatigue is of great importance for the patient. Despite affecting the patients' lives to this extent, fatigue and discomfort have often been overlooked and neglected symptoms due to their subjective nature. Various pharmacological and non-pharmacological treatment methods are used to control fatigue due to CRF or HD and to bring the desired patient comfort. One of the non-pharmacological methods is massage. Massage can be defined as scientific systematic manipulations applied to body tissues in order to affect the locomotor system and nervous system as well as the general circulation. There are studies in the literature where various applications are applied to HD patients to affect fatigue and comfort. However, it is striking that there is no study examining the effect of massage on the comfort and fatigue levels of patients receiving HD treatment. Therefore, the research was planned to examine the effect of massage on the comfort level and fatigue level of HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being 18 years of age or older
* Receiving hemodialysis treatment in a dialysis unit for at least six months
* Not having a condition that prevents verbal communication
* Not having a psychiatric problem

Exclusion Criteria:

* Patients who left the study at any stage
* Patients who had been receiving hemodialysis treatment for less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hemodialysis Comfort Scale | Up to 4 weeks
  The scale developed by Sahin Orak and his colleagues in 2017 consists of nine items and two sub-dimensions. These sub-dimensions are; "Relaxation" (7-9) and "Overcoming" (1- 6). The scale is a five-point Likert type (1: never -5: always). Items 1-3 and 5-9 of the scale are reverse coded. The lowest score that can be obtained from the scale is 9, the highest score is 45. The higher the score, the higher the comfort level.
Piper Fatigue Scale | Up to 4 weeks
  The scale was developed by Barbara F. Piper and her friends in 1987 and adapted to Turkish by Can and her friends in 2001. The scale consists of 22 items and four sub-dimensions. These are; "Behavior/Violence" (2-7); "Affect" (8-12), "Sensory" (5 items; 13-17) and "Cognitive/Psychological" (18-23). In addition to this, there are five items (1 and 24-27) that are not used in calculating the fatigue score, but are recommended to remain in the scale because they are important in evaluating data related to fatigue. The scale is evaluated using a 0-10 Vizuel Analog Scale. The total score obtained from the scale is divided by the number of items. The minimum score that can be obtained from the scale is 0, and the maximum score is 10. The higher the score, the more fatigue the individual feels.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No